CLINICAL TRIAL: NCT02602535
Title: Mindfulness-Oriented Recovery Enhancement For Chronic Pain and Prescription Opioid Misuse in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00078615
Record Dates: First submitted 2015-10-26; First posted 2015-11-11 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain; Opioid Use Disorders
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- M.O.R.E. (Experimental): Participants will attend a Mindfulness-Oriented Recovery Enhancement (MORE) group weekly for eight weeks.
  Interventions: Behavioral: Mindfulness-Oriented Recovery Enhancement
- Support Group (Active Comparator): Participants will attend a support group weekly for eight weeks.
  Interventions: Behavioral: Support Group

INTERVENTIONS:
Behavioral: Mindfulness-Oriented Recovery Enhancement — Mindfulness-Oriented Recovery Enhancement (MORE) is a group behavioral intervention that unites mindfulness training, cognitive reappraisal, and positive psychological principles into an integrative intervention strategy targeting mechanisms of pain and opioid misuse.
  Arms: M.O.R.E.
Behavioral: Support Group — A conventional support group will allow participants to express emotions, share experiences, and receive social support under the guidance of a skilled therapist.
  Arms: Support Group

SUMMARY:
The central aim of this study is to test the efficacy of Mindfulness-Oriented Recovery Enhancement (MORE), an intervention designed to disrupt the risk chain leading from chronic pain to prescription opioid misuse and addiction. The investigators plan to conduct a full scale clinical trial to determine whether MORE (relative to a support group control condition) can reduce symptoms of chronic pain and opioid misuse among patients who are receiving pain management in primary care via long-term opioid analgesic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60+
* Current back pain diagnosis as determined from ICD-9 codes in claims data (including but not limited to ICD-9 diagnoses 724.x, or 847.x) or current chronic pain diagnosis determined by physician assessment (including but not limited to ICD-9 diagnoses 338.0, 338.21, 338.22, 338.28, 338.29, 338.4)
* Current use of prescription opioid agonist or mixed agonist-antagonist analgesics for >90 days, and evidence of opioid misuse as indicated by the Current Opioid Misuse Measure
* Willingness to participate in study interventions and assessments

Exclusion Criteria:

* Prior experience with Mindfulness-Based Stress Reduction, Mindfulness-Based Cognitive Therapy, or Mindfulness-Based Relapse Prevention
* Active suicidality, schizophrenia, psychotic disorder, and/or substance dependence (other than opioid dependence)
* Presence of clinically unstable systemic illness judged to interfere with treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-01; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in opioid misuse | Change from baseline through study completion (9 months post-treatment)
  Opioid misuse as evidenced by triangulated aggregate of Current Opioid Misuse Measure and/or clinician assessment via Addiction Behaviors Checklist and/or urine screen
Change in pain severity and interference | Change from baseline through study completion (9 months post-treatment)
  Brief Pain Inventory

SECONDARY OUTCOMES:
Change in opioid craving | Change from baseline through study completion (9 months post-treatment)
  Opioid craving measure from Wasan et al. 2012
Change in psychological distress | Change from baseline through study completion (9 months post-treatment)
  Depression Anxiety Stress Scale
Change in opioid dose | Change from baseline through study completion (9 months post-treatment)
  Opioid dose converted into morphine equivalents via standardized equianalgesic tables

OTHER OUTCOMES:
Change in nonreactivity | Change from baseline through post-treatment (8 weeks from beginning of treatment)
  subscale on Five Facet Mindfulness Questionnaire
Change in interoceptive awareness | Change from baseline through post-treatment (8 weeks from beginning of treatment)
  Interoceptive awareness as evidenced by the Multidimensional Assessment of Interoceptive Awareness
Change in reinterpretation of pain sensations | Change from baseline through post-treatment (8 weeks from beginning of treatment)
  Reinterpretation of pain sensations subscale on the Coping Strategies Questionnaire
Change in emotion regulation | Change from baseline through post-treatment (8 weeks from beginning of treatment)
  Emotion regulation as evidenced by responses on the Emotion Regulation Task
Change in positive emotion | Change from baseline through post-treatment (8 weeks from beginning of treatment)
  Positive emotion as evidenced by the PANAS
Change in cue-reactivity | Change from baseline through post-treatment (8 weeks from beginning of treatment)
  Cue-reactivity as evidenced by attentional bias and central-autonomic responses during cue-exposure
Change in attention to positive information | Change from baseline through post-treatment (8 weeks from beginning of treatment)
  Attention to positive information as evidenced by the APNIS
Change in anhedonia | Change from baseline through study completion (9 months post-treatment)
  Anhedonia as evidenced by the Snaith Hamilton Anhedonia and Pleasure Scale (SHAPS), from 14 to 56, with lower scores meaning less anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garland, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Primary Care Clinics, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Garland EL, Hudak J, Hanley AW, Bernat E, Froeliger B. Positive Emotion Dysregulation in Opioid Use Disorder and Normalization by Mindfulness-Oriented Recovery Enhancement: A Secondary Analysis of a Randomized Clinical Trial. JAMA Psychiatry. 2025 Jul 1;82(7):654-662. doi: 10.1001/jamapsychiatry.2025.0569. PMID 40305010
- [Derived] Garland EL, Hanley AW, Nakamura Y, Barrett JW, Baker AK, Reese SE, Riquino MR, Froeliger B, Donaldson GW. Mindfulness-Oriented Recovery Enhancement vs Supportive Group Therapy for Co-occurring Opioid Misuse and Chronic Pain in Primary Care: A Randomized Clinical Trial. JAMA Intern Med. 2022 Apr 1;182(4):407-417. doi: 10.1001/jamainternmed.2022.0033. PMID 35226053

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT02602535/SAP_000.pdf